CLINICAL TRIAL: NCT00152776
Title: Treatment of Climacteric Symptoms With Ovaria Comp - A Prospective Randomized Placebo Controlled Doubleblind Study
Brief Title: Treating Climacteric Symptoms With a Complex Homeopathic Remedy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Wala GmbH (Industry)
Responsible Party: Principal Investigator, Cornelia von Hagens, Principal Investigator, Heidelberg University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD04
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Menopause; Anxiety Disorders; Depression
Keywords: menopausal symptoms; complementary medicine
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I (Placebo Comparator): ovaria comp 10 Globuli 3 times per day 24 weeks - Placebo 12 weeks
  Interventions: Drug: ovaria comp 10 globuli 3 times per day 24 weeks
- Group II (Placebo Comparator): Placebo 12 weeks - ovaria comp 10 globuli 3 times per day 24 weeks
  Interventions: Drug: ovaria comp 10 globuli 3 times per day 24 weeks
- Group III (Placebo Comparator): ovaria comp 10 globuli 3 times per day 12 weeks - Placebo 12 weeks - ovaria comp 10 globuli 3 times per day 12 weeks
  Interventions: Drug: ovaria comp 10 globuli 3 times per day 24 weeks

INTERVENTIONS:
Drug: ovaria comp 10 globuli 3 times per day 24 weeks — order of intervention and placebo varies between Groups I-III
  Other Names: placebo globuli 3 times per day 12 weeks

SUMMARY:
The purpose of this study is to determine whether ovaria comp. is effective in relieving climacteric symptoms.

DETAILED DESCRIPTION:
Complementary treatments for climacteric symptoms are used by many women although their efficacy and safety is mostly unproven.

The use of the complex homeopathic remedy Ovaria comp. for the relief of climacteric symptoms will be examined in this three-armed intervention trial and measured with the menopause rating scale II before and after each study phase of 12 weeks. Participants will receive the verum during two treatment phases of 12 weeks and the placebo during one treatment phase of 12 weeks in different sequences and are stratified for post- and perimenopausal status.

ELIGIBILITY:
Inclusion Criteria:

* Climacteric symptoms>=3 Points in Menopause Rating Scale (MRS) II
* Communication possible

Exclusion Criteria:

* Hormone replacement therapy within 2 weeks prior to study inclusion
* Other complementary treatments 7 days before and during the study
* Climacteric symptoms caused by operation, chemotherapy or hormonal therapy of cancer
* Allergy to components of the remedy, especially bee poison

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Climacteric symptoms | 12 weeks
  sum score of the menopause rating scale (MRS II) before and after 12 weeks of treatment

SECONDARY OUTCOMES:
Climacteric symptoms (vegetative, psychological, urogenital subscales of the MRS II) | 12 weeks
  difference of the subscales of the menopause rating scale before and after 12 weeks of treatment
Follow-up for another 12 weeks of treatment or after cross-over to the placebo group | 12+12 weeks
  sum score and subscales of the MRS II
Follow-up for cross-over to placebo after 24 weeks of treatment | 12+12+12 weeks
  sum score and subscales of the MRS II
Diurnal profile of cortisol level before and after treatment phases | 12+12+12 weeks
  cortisol (saliva: morning, noon, evening)
Anxiety and depression measured by Hospital Anxiety and Depression Scale (HADS-D) before and after treatment period | 12+12+12 weeks
  Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia U von Hagens, MD, Principal Investigator — Heidelberg University
Locations (1):
- Department of Complementary and Integrative Medicine, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] von Hagens C, Schiller P, Godbillon B, Osburg J, Klose C, Limprecht R, Strowitzki T. Treating menopausal symptoms with a complex remedy or placebo: a randomized controlled trial. Climacteric. 2012 Aug;15(4):358-67. doi: 10.3109/13697137.2011.597895. Epub 2011 Oct 23. PMID 22017387